CLINICAL TRIAL: NCT04545268
Title: Prehabilitation for Cardiac Surgery in Patients With Reduced Exercise Tolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Andrey Bezdenezhnykh, Senior Researcher of Comorbidity in Cardiovascular Diseases Laboratory, PhD, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020_4_19_32
Record Dates: First submitted 2020-08-18; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Sarcopenia; Exercise Intolerance; Heart Failure; Peripheral Artery Disease
MeSH Terms: conditions — Sarcopenia; Heart Failure; Peripheral Arterial Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This is a single-blinded, randomized controlled longitudinal study design to determine if NMES will increase muscle mass and strength and improve exercise capacity thus improving likelihood of engagement with a structured exercise program. Patients will be randomized to either intervention that includes NMES or to a sham control group. In order to ensure that the two groups are comparable between treatment and sham interventions, the participants will be randomized according to gender. Randomization via minimization will be used in order to avoid an unbalanced number of women in the two comparison groups due to chance. A file of the computer-generated random assignments will be kept.
Who Masked: Outcomes Assessor
Masking Description: The Investigator will collect baseline data before the participant is randomized. The intervention/sham will be set-up by the Investigator. The Investigator who is trained in both NMES and Sham intervention will then look at the randomization schedule and set up and train the participants on equipment use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator)
  Interventions: Device: Transcutaneous electrical stimulation
- NMES group (Experimental)
  Interventions: Device: Neuromuscular electrical stimulation (NMES)

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) — NMES will carried out with four-channel myostimulator "Beurer EM80" (Germany). Self-adhesive electrodes locates above the quadriceps, the duration of the NMES session was 60 minutes, including 5-minute periods of heating and hitch. Throughout the series, rectangular pulses with a frequency of 45 Hz will modulate. As a result, tonic contraction of these muscles will induce for 12 seconds, followed by a pause of 5 seconds. The amplitude of electrical exposure will select separately for each of the four channels until good muscle contraction (visually or by palpation) without pain. Electrical stimulation will start from the second day after the admission to preoperative department and will carried out during the entire preoperative period (about 10 days).
  Arms: NMES group
Device: Transcutaneous electrical stimulation — For the Sham group, electrodes will follow the same site, but the stimulation will only increase to an intermittent tingling sensation with the machine setting on TENS instead of NMES which is not enough to make noticeable changes in muscle mass or circulation. Intensity settings will not change over time.
  Arms: Control group

SUMMARY:
Among patients awaiting cardiac surgery, a significant proportion are patients with severe angina, heart failure (HF) and peripheral atherosclerosis. These factors are predictors of an unfavorable near and long-term prognosis after open cardiac surgery. It is known that the restriction of motor activity in patients with peripheral atherosclerosis and HF leads to loss of muscle mass, as well as to a decrease in its strength and endurance: secondary (disuse) sarcopenia is formed. In patients with peripheral atherosclerosis and HF, the low functional status of skeletal muscles is associated with a poor prognosis, regardless of gender, age, and concomitant coronary artery disease. A number of studies have shown that the deterioration of muscle status before abdominal, orthopedic and vascular surgery interferes with the close results of surgery, increases the number of complications, the length of ICU and in-hospital stay. Thus, sarcopenia serves as an additional factor worsening the prognosis. Therefore, efforts aimed at improving the functional status in patients planning an open cardiosurgical surgery seem to be very justified.

Standard preoperative management of patients includes the identification and correction of comorbidities and the optimal medical treatment. The idea of "rehabilitation" means an additional improvement in the functional capabilities of patients awaiting surgery. Prevention includes outpatient outreach and educational work by nurses, as well as preoperative physical exercises. For this, multi-level training is used: respiratory exercises for the patients with the most severe illness, free movements of the limbs without load, or bike or treadmill training with increasing load for tolerable patients.

However, adequate physical rehabilitation is difficult particularly on an outpatient basis. Low adherence is due in part to inadequate strength and inability to tolerate or sustain even low levels of activity due to angina, chronic lower limb ischemia and heart failure symptoms.

In this study, the investigators propose to use neuromuscular electrical stimulation (NMES) to assist patient initiation of quadriceps strengthening in order to progressively increase low exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting for elective cardiovascular procedure (CABG, valvular or thoracic aorta) unable to walk more than 300 meters during six-minuite walking test due to angina, dyspnea or limb ischemia
* no weakness of lower limbs
* stable hemodynamic, already received standard treatment based on patient condition
* able to follow protocol procedures
* assigned the informed consent
* do not regularly exercise (10 minutes or more a day of exercise most days of the week for the past week).

Exclusion Criteria:

* urgent indications for surgery or counterindication for elective operation
* already receive NMES at femoris area in last 6 weeks before admission
* Patients, who have undertaken cardiac rehab within the 12 months prior to enrollment
* Cognitive, orthopedic or neurological disorders or other impairment which prevents accurate application of intervention or inability to provide informed consent
* End Stage Renal Disease
* Uncontrolled arrhythmia's or 3rd degree AV heart block
* Those with wounds over area of proper placement of electrodes

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in strength test (Dynamometer) from baseline to post EMS in EMS vs. controls | From baseline to post EMS (at least 6th day after baseline)
  Strength Assessment using a portable hand-held dynamometer (Lafayette Manual Muscle Test System 001165)
Change in strength test (Dynamometer) from post EMS to pre-discharge in EMS vs. controls | from post EMS (at least 6th day after baseline) to the end of hospitalisation (expected an average of 10 days)
  Strength Assessment will be done using a portable hand-held dynamometer (Lafayette Manual Muscle Test System 001165).

SECONDARY OUTCOMES:
Change in 6-minute walk test distance from baseline to post EMS in EMS vs. controls | Baseline, post EMS (at least 6th day after baseline)
  Participants will be instructed to move as quickly as they feel safe and comfortable over the 50-meter course for 6 minutes. As per the protocol, participants will be allowed to stop and rest if necessary
Change in 6-minute walk test distance from post EMS to pre-discharge in EMS vs. controls | Baseline, post EMS (at least 6th day after baseline)
  Participants will be instructed to move as quickly as they feel safe and comfortable over the 50-meter course for 6 minutes. As per the protocol, participants will be allowed to stop and rest if necessary

OTHER OUTCOMES:
Change in length of stay (LOS) in ICU in EMS vs. controls. | From the end of cardiac procedure to the end of ICU stay (expected an average of 1 day)
Change in length of stay (LOS) in postoperative department in EMS vs. controls | From the end of cardiac procedure to the end of hospitalisation (expected an average of 10 days)
  number of days
Change in mechanical ventilation duration in EMS vs. controls | from the intubation to the extubation (expected an average of 7 hours)
  number of minuits
Rate of postoperative complication or death | From the end of cardiac procedure to the end of hospitalisation (expected an average of 10 days)
  Any complication wich required hospitalisation prolongation or additional procedures (eg pleural or pericardial punction, renal replacemen therapy, pneumonia, wound complications etc.) or death

CONTACTS AND LOCATIONS:
Overall Officials: Andrey V Bezdenezhnykh, PhD, Principal Investigator — Research Institute for Complex Issues of Cardiovacular Diseases
Locations (1):
- Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo, Russia

IPD SHARING:
Plan to Share IPD: No